CLINICAL TRIAL: NCT02453126
Title: Fibrostenotic Eosinophilic Esophagitis: Endoscopic, Histologic and Molecular Characterization and Evaluation of Clinical Assessment Tools
Brief Title: Fibrostenotic Eosinophilic Esophagitis: Assessment Tools
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0594; UL1TR001082 (NIH)
Record Dates: First submitted 2014-09-16; First posted 2015-05-25 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Esophageal Stricture
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophageal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol addresses a central hypothesis that fibrostenotic Eosinophilic Esophagitis (EoE) is characterized by abnormal esophageal structure and compliance compared to non fibrostenotic EoE and that distinctive cellular and molecular profiles predict the fibrostenotic phenotype. This study aims to define and assess the changes that occur in the structure and dynamics of the esophageal wall in pediatric Eosinophilic Esophagitis along with characterizing the histologic and molecular patterns in fibrostenotic EoE.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a clinical upper endoscopy with biopsy

Exclusion Criteria:

* Known connective tissue disorder
* Increased risk of bleeding
* Inflammatory bowel disease, celiac disease, eosinophilic gastroenteritis, or any autoimmune disease
* Other esophageal disease including known achalasia; history of caustic ingestion, esophageal surgery esophageal stricture for other known reason or other esophageal injury.
* Use of oral or intravenous steroids in the preceding 60 days. (Swallowed topical fluticasone, budesonide, etc not included as exclusion criteria.)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, ages 5 to 18 years, scheduled to undergo a clinical upper endoscopy with biopsy for suspected or confirmed Eosinophilic Esophagitis.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-12; Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Stricture, as measured by endoscopic assessment | Day 1

SECONDARY OUTCOMES:
Decreased esophageal distensibility, as determined by EndoFlip | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Calies Menard-Katcher, MD, Principal Investigator — University of Colorado/Childrens Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States